CLINICAL TRIAL: NCT03982199
Title: A Randomized, Double-blind, Placebo-controlled Phase 2b Study to Assess the Efficacy, Immunogenicity and Safety of an Ad26.RSV.preF-based Regimen in the Prevention of RT PCR-confirmed RSV-mediated Lower Respiratory Tract Disease in Adults Aged 65 Years and Older
Brief Title: A Study of an Ad26.RSV.preF-based Regimen in the Prevention of Reverse Transcriptase Polymerase Chain Reaction (RT-PCR)-Confirmed Respiratory Syncytial Virus (RSV)-Mediated Lower Respiratory Tract Disease in Adults Aged 65 Years and Older
Acronym: CYPRESS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated early by the sponsor due to strategic reprioritization reasons.
Sponsor: Janssen Vaccines & Prevention B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CR108634; VAC18193RSV2001 (Other: Janssen Vaccines & Prevention B.V.)
Record Dates: First submitted 2019-06-10; First posted 2019-06-11 (Actual); Results first posted 2023-07-24 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Respiratory Syncytial Viruses; Respiratory Tract Diseases
MeSH Terms: conditions — Respiratory Tract Diseases | interventions — Respiratory Syncytial Virus Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1: RSV Vaccine (Experimental): Participants will receive a single intramuscular (IM) injection of an adenovirus serotype 26 (Ad26)-based respiratory syncytial virus (RSV) vaccine at a single dose level on Day 1. Participants will then be divided into revaccination subcohorts: 1A, 1B, and 1C to receive revaccination with Ad26.RSV.preF based vaccine at 1 year, 2 years, and 3 years respectively after the first vaccination.
  Interventions: Biological: RSV Vaccine
- Group 2: Placebo (Placebo Comparator): Participants will receive a single IM injection of placebo control on Day 1. Participants will then be divided into revaccination subcohorts 2A, 2B, and 2C, and will first receive Ad26.RSV.preF based vaccine at years 1, 2, and 3. In subcohorts 2A and 2B, participants will receive a revaccination one year later with either Ad26.RSV.preF based vaccine, study vaccine A or study vaccine B.
  Interventions: Biological: RSV Vaccine; Biological: Placebo

INTERVENTIONS:
Biological: RSV Vaccine — Participants will receive a single IM injection of an Ad26-based RSV vaccine at a single dose level on Day 1 and revaccination after either 1 year, 2 years, or 3 years.
Biological: Placebo — Participants will receive a single IM injection of placebo control on Day 1.
  Arms: Group 2: Placebo

SUMMARY:
The purpose of this study is to demonstrate the efficacy of active study vaccine in the prevention of reverse transcriptase polymerase chain reaction (RT-PCR) confirmed respiratory syncytial virus (RSV)-mediated lower respiratory tract disease (LRTD), when compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have a body mass index (BMI) less than (<)40 kilogram per meter square (kg/m^2)
* Before randomization, a woman must be: postmenopausal (postmenopausal state is defined as no menses for 12 months without an alternative medical cause); and not intending to conceive by any methods
* Participant must be either in good or stable health. Participants may have mild to moderate underlying illnesses such as chronic cardiac diseases and chronic lung disease (asthma and chronic obstructive pulmonary disease [COPD]), congestive heart failure (CHF), hypertension, type 2 diabetes mellitus, hyperlipoproteinemia, or hypothyroidism, as long as their symptoms and signs are stable and medically controlled in the judgment of the investigator. Participants will be included on the basis of physical examination, medical history, and vital signs performed between informed consent form (ICF) signature and vaccination on Day 1
* From the time of vaccination through 3 months after vaccination, participant agrees not to donate blood
* Participant must be able to read, understand, and complete questionnaires in the eDiary (or a paper safety diary, if designated by the sponsor)
* Participant must be willing to provide verifiable identification, have means to be contacted and to contact the investigator during the study

Exclusion Criteria:

* Participant has an acute illness (including acute respiratory illnesses) or body temperature greater than or equal to (>=)38.0 degree Celsius (ºC) within 24 hours prior to administration of study vaccine. In such a situation, enrollment at a later date is permitted
* Participant has a severe or potentially life-threatening chronic disorder such as severe chronic cardiac diseases and severe chronic lung disease (asthma and COPD), advanced CHF, end-stage renal disease with or without dialysis, clinically unstable cardiac disease, Alzheimer's disease, or has any condition for which, in the opinion of the investigator, participation would not be in the best interest of the participant (example: compromise well-being) or that could prevent, limit, or confound the protocol-specified assessments
* Participant has a history of malignancy within 5 years before screening (exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, or malignancy, which is considered cured with minimal risk of recurrence)
* Per medical history, participant has chronic active hepatitis B or hepatitis C infection
* Per medical history, participant has human immunodeficiency virus (HIV) type 1 or type 2 infection
* Participant has a known allergy, or history of anaphylaxis or other serious adverse reactions to vaccines or vaccine components (including any of the constituents of the study vaccine)

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 5815 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2022-06-06 (Actual); Study Completion 2023-05-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Vaccines & Prevention B.V. Clinical Trial, Study Director — Janssen Vaccines & Prevention B.V.
Locations (40):
- United States (40):
  - Optimal Research, Huntsville, Alabama
  - Synexus Clinical Research US Inc, Chandler, Arizona
  - Synexus Clinical Research US Inc, Phoenix, Arizona
  - Central Phoenix Medical Clinic, Phoenix, Arizona
  - Anaheim Clinical Trials, LLC, Anaheim, California
  - Paradigm Clinical Research Centers, Inc., Redding, California
  - Benchmark Research, Sacramento, California
  - Optimal Research, San Diego, California
  - Synexus Clinical Research US Inc, Aurora, Colorado
  - Lynn Institute, Colorado Springs, Colorado
  - Optimal Research, Melbourne, Florida
  - Advanced Clinical Research, Boise, Idaho
  - Optimal Research, Peoria, Illinois
  - Synexus Clinical Research US Inc, Evansville, Indiana
  - The Iowa Clinic, West Des Moines, Iowa
  - Hutchinson Clinic, Hutchinson, Kansas
  - Johnson County Clin-Trials, Lenexa, Kansas
  - Heartland Research Associates, LLC, Newton, Kansas
  - Heartland Research Associates, LLC, Wichita, Kansas
  - Optimal Research, Rockville, Maryland
  - Synexus Clinical Research US Inc, Richfield, Minnesota
  - The Center For Pharmaceutical Research, Kansas City, Missouri
  - Sundance Clinical Research, St Louis, Missouri
  - Synexus Clinical Research US Inc, St Louis, Missouri
  - Synexus Clinical Research US Inc, Elkhorn, Nebraska
  - Synexus Clinical Research US Inc, Omaha, Nebraska
  - United Medical Associates, Binghamton, New York
  - Regional Clinical Research, Inc., Endwell, New York
  - University of Rochester / Rochester General Hospital, Rochester, New York
  - Synexus Clinical Research US Inc, Akron, Ohio
  - Synexus Clinical Research US Inc, Cincinnati, Ohio
  - Rapid Medical Research, Cleveland, Ohio
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Omega Medical Research, Warwick, Rhode Island
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - Optimal Research, Austin, Texas
  - Ventavia Research Group, LLC, Fort Worth, Texas
  - Synexus Clinical Research US Inc, Murray, Utah
  - Advanced Clinical Research, Salt Lake City, Utah
  - Advanced Clinical Research, West Jordan, Utah

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency.
  As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] Falsey AR, Hosman T, Bastian AR, Vandenberghe S, Chan EKH, Douoguih M, Heijnen E, Comeaux CA, Callendret B; CYPRESS investigators. Long-term efficacy and immunogenicity of Ad26.RSV.preF-RSV preF protein vaccine (CYPRESS): a randomised, double-blind, placebo-controlled, phase 2b study. Lancet Infect Dis. 2024 Sep;24(9):1015-1024. doi: 10.1016/S1473-3099(24)00226-3. Epub 2024 May 24. PMID 38801826
- [Derived] Falsey AR, Williams K, Gymnopoulou E, Bart S, Ervin J, Bastian AR, Menten J, De Paepe E, Vandenberghe S, Chan EKH, Sadoff J, Douoguih M, Callendret B, Comeaux CA, Heijnen E; CYPRESS Investigators. Efficacy and Safety of an Ad26.RSV.preF-RSV preF Protein Vaccine in Older Adults. N Engl J Med. 2023 Feb 16;388(7):609-620. doi: 10.1056/NEJMoa2207566. PMID 36791161

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants in the main cohort who did not enter the re-vaccination subcohorts continued in the main cohort up to Day 1095. Hence, the assessments for both main cohorts and re-vaccination subcohorts were conducted in parallel until Day 1095 (end of main cohort).
Groups:
- Arm 1: Main Cohort: Group 1: Ad26.RSV.preF and RSV preF Protein (Protein Mixture): Adult participants aged greater than or equal to (>=) 65 years received a single intramuscular (IM) injection of adenovirus serotype 26 respiratory syncytial virus pre-fusion conformation stabilized F-protein (Ad26.RSV.preF) 1*10^11 viral particles (vp) and RSV preF protein 150 micrograms (mcg) (protein mixture) on Day 1. Participants were divided into revaccination subcohorts: 1A, 1B, and 1C. Participants further received revaccination with the Ad26.RSV.preF 1*10^11 vp and RSV preF protein 150 mcg (protein mixture) at 1 (Subcohort 1A), 2 (Subcohort 1B), and 3 (Subcohort 1C) years, respectively after the first vaccination on Day 1. Participants who were not re-vaccinated continued in the main cohort and were followed up for safety assessments until Day 1095.
- Arm 2: Main Cohort: Group 2: Placebo: Adult participants aged >=65 years received a single IM injection of placebo on Day 1. Participants were divided into revaccination subcohorts: 2A, 2B, and 2C. Participants further received revaccination with Ad26.RSV.preF 1*10^11 vp and RSV preF protein 150 mcg (protein mixture) at 1 (Subcohort 2A), 2 (Subcohort 2B), and 3 (Subcohort 2C) years, respectively after the first vaccination on Day 1. Participants in subcohorts 2A and 2B were additionally re-randomised in three groups at Year 3 and Year 4, respectively, to receive either Ad26.RSV.preF 1*10^11 vp alone, RSV preF protein 150 mcg alone or the Ad26.RSV.preF 1*10^11 vp and RSV preF protein 150 mcg (protein mixture). Participants who were not re-vaccinated continued in the main cohort and were followed up for safety assessments until Day 1095.
- Arm 3: Revaccination (ReVacc) Subcohort 1A: Ad26.RSV.preF/RSV preF Protein (Protein Mixture): Eligible participants who received IM injection of Ad26.RSV.preF 1*10^11 vp and RSV preF protein 150 mcg (protein mixture) on Day 1 in the main cohort entered the revaccination subcohort 1A and received IM injection of the protein mixture at the same dose level on Day 365. Participants were then followed up for safety assessments till Day 730.
- Arm 4: ReVacc Subcohort 2A: Placebo to Ad26.RSV.preF/RSV preF Protein Mixture: Eligible participants who received IM injection of placebo on Day 1 in the main study cohort entered the revaccination subcohort and received Ad26.RSV.preF 1*10^11 vp and RSV preF protein 150 mcg (protein mixture) on Day 365. Participants were then followed up for safety assessments till Day 730.
- Arm 5: ReVacc Subcohort 2A: Placebo to Ad26.RSV.preF/RSV preF Protein + Ad26.RSV.PreF Alone: Eligible participants who received IM injection of placebo on Day 1 in the main cohort followed by Ad26.RSV.preF 1*10^11 vp and RSV preF protein 150 mcg (protein mixture) on Day 365 in the revaccination subcohort further received Ad26.RSV.preF 1*10^11 vp alone as IM injection on Day 730. Participants were then followed up for safety assessments till Day 1095.
- Arm 6: ReVacc Subcohort 2A: Placebo to Ad26.RSV.preF/RSV preF Protein + RSV preF Protein Alone: Eligible participants who received IM injection of placebo on Day 1 in the main cohort followed by Ad26.RSV.preF 1*10^11 vp and RSV preF protein (protein mixture) on Day 365 in the revaccination subcohort further received RSV preF protein 150 mcg alone as IM injection on Day 730. Participants were then followed up for safety assessments till Day 1095.
- Arm 7: ReVacc Subcohort 2A: Placebo to Ad26.RSV.preF/RSV preF Protein (Protein Mixture): Eligible participants who received IM injection of placebo on Day 1 in the main study cohort entered the revaccination subcohort and received IM injection of Ad26.RSV.preF 1*10^11 vp and RSV preF protein 150 mcg (protein mixture) on Day 365 and 730. Participants were then followed up for safety assessments till Day 1095.
- Arm 8: ReVacc Subcohort 1B: Ad26.RSV.preF/RSV preF Protein (Protein Mixture): Eligible participants who received IM injection of Ad26.RSV.preF 1*10^11 vp and RSV preF protein 150 mcg (protein mixture) on Day 1 in the main cohort entered the revaccination subcohort and received the protein mixture at the same dose level on Day 730. Participants were then followed up for safety assessments till Day 1095.
- Arm 9: ReVacc Subcohort 2B:Placebo to Ad26.RSV.preF/RSV preF Protein (Protein Mixture): Eligible participants who received IM injection of placebo on Day 1 in the main cohort entered the revaccination subcohort and received IM injection of Ad26.RSV.preF 1*10^11 vp and RSV preF protein 150 mcg (protein mixture) on Day 730. Participants were then followed up for safety assessments till Day 1095.
- Arm 10: ReVacc Subcohort 2B: Placebo to Ad26.RSV.preF/RSV preF Protein + Ad26.RSV.preF: Eligible participants who received IM injection of placebo on Day 1 in the main cohort entered the revaccination subcohort and received IM injection of Ad26.RSV.preF 1*10^11 vp and RSV preF protein 150 mcg (protein mixture) on Day 730 followed by Ad26.RSV.preF 1*10^11 vp alone on Day 1095. Participants were then followed up for safety assessments till Day 1460.
- Arm 11: ReVacc Subcohort 2B: Placebo to Ad26.RSV.preF/RSV preF Protein + RSV preF Protein Alone: Eligible participants who received IM injection of placebo on Day 1 in the main cohort entered the revaccination subcohort and received IM injection Ad26.RSV.preF 1*10^11 vp and RSV preF protein 150 mcg (protein mixture) on Day 730 followed by RSV preF protein 150 mcg alone on Day 1095. Participants were then followed up for safety assessments till Day 1460.
- Arm 12: ReVacc Subcohort 2B: Placebo to Ad26.RSV.preF/RSV preF Protein (Protein Mixture): Eligible participants who received IM injection of placebo on Day 1 in the main cohort entered the revaccination subcohort and received IM injection of Ad26.RSV.preF 1*10^11 vp and RSV preF protein 150 mcg (protein mixture) on Days 730 and Day 1095. Participants were then followed up for safety assessments till Day 1460.
- Arm 13: ReVacc Subcohort 1C: Ad26.RSV.preF/RSV preF Protein (Protein Mixture): Eligible participants who received IM injection of Ad26.RSV.preF 1*10^11 vp and RSV preF protein 150 mcg (protein mixture) on Day 1 in the main cohort entered the revaccination subcohort and received the protein mixture at the same dose level on Day 1095. Participants were then followed up for safety assessments till Day 1460.
- Arm 14: ReVacc Subcohort 2C: Placebo to Ad26.RSV.preF/RSV preF Protein (Protein Mixture): Eligible participants who received IM injection of placebo on Day 1 in the main cohort entered the revaccination subcohort and received IM injection of Ad26.RSV.preF 1*10^11 vp and RSV preF protein 150 mcg (protein mixture) on Day 1095. Participants were then followed up for safety assessments till Day 1460.
Period: Main Cohorts (Day 1 up to Day 1095)
Arm/Group | Arm 1: Main Cohort: Group 1: Ad26.RSV.preF and RSV preF Protein (Protein Mixture) | Arm 2: Main Cohort: Group 2: Placebo | Arm 3: Revaccination (ReVacc) Subcohort 1A: Ad26.RSV.preF/RSV preF Protein (Protein Mixture) | Arm 4: ReVacc Subcohort 2A: Placebo to Ad26.RSV.preF/RSV preF Protein Mixture | Arm 5: ReVacc Subcohort 2A: Placebo to Ad26.RSV.preF/RSV preF Protein + Ad26.RSV.PreF Alone | Arm 6: ReVacc Subcohort 2A: Placebo to Ad26.RSV.preF/RSV preF Protein + RSV preF Protein Alone | Arm 7: ReVacc Subcohort 2A: Placebo to Ad26.RSV.preF/RSV preF Protein (Protein Mixture) | Arm 8: ReVacc Subcohort 1B: Ad26.RSV.preF/RSV preF Protein (Protein Mixture) | Arm 9: ReVacc Subcohort 2B:Placebo to Ad26.RSV.preF/RSV preF Protein (Protein Mixture) | Arm 10: ReVacc Subcohort 2B: Placebo to Ad26.RSV.preF/RSV preF Protein + Ad26.RSV.preF | Arm 11: ReVacc Subcohort 2B: Placebo to Ad26.RSV.preF/RSV preF Protein + RSV preF Protein Alone | Arm 12: ReVacc Subcohort 2B: Placebo to Ad26.RSV.preF/RSV preF Protein (Protein Mixture) | Arm 13: ReVacc Subcohort 1C: Ad26.RSV.preF/RSV preF Protein (Protein Mixture) | Arm 14: ReVacc Subcohort 2C: Placebo to Ad26.RSV.preF/RSV preF Protein (Protein Mixture)
Started | 2909 | 2906 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaccinated | 2891 | 2891 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 1875 | 1897 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 1034 | 1009 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 152 | 159 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 39 | 33 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 514 | 503 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 12 | 14 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Technical Problems | 10 | 8 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 39 | 38 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Site terminated by Sponsor | 26 | 21 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Study Terminated by Sponsor | 129 | 117 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 80 | 83 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Randomized but not vaccinated | 18 | 15 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 4 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Initiated prohibited medication | 11 | 11 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Revacc Subcohorts (From Day 365 to 730)
Arm/Group | Arm 1: Main Cohort: Group 1: Ad26.RSV.preF and RSV preF Protein (Protein Mixture) | Arm 2: Main Cohort: Group 2: Placebo | Arm 3: Revaccination (ReVacc) Subcohort 1A: Ad26.RSV.preF/RSV preF Protein (Protein Mixture) | Arm 4: ReVacc Subcohort 2A: Placebo to Ad26.RSV.preF/RSV preF Protein Mixture | Arm 5: ReVacc Subcohort 2A: Placebo to Ad26.RSV.preF/RSV preF Protein + Ad26.RSV.PreF Alone | Arm 6: ReVacc Subcohort 2A: Placebo to Ad26.RSV.preF/RSV preF Protein + RSV preF Protein Alone | Arm 7: ReVacc Subcohort 2A: Placebo to Ad26.RSV.preF/RSV preF Protein (Protein Mixture) | Arm 8: ReVacc Subcohort 1B: Ad26.RSV.preF/RSV preF Protein (Protein Mixture) | Arm 9: ReVacc Subcohort 2B:Placebo to Ad26.RSV.preF/RSV preF Protein (Protein Mixture) | Arm 10: ReVacc Subcohort 2B: Placebo to Ad26.RSV.preF/RSV preF Protein + Ad26.RSV.preF | Arm 11: ReVacc Subcohort 2B: Placebo to Ad26.RSV.preF/RSV preF Protein + RSV preF Protein Alone | Arm 12: ReVacc Subcohort 2B: Placebo to Ad26.RSV.preF/RSV preF Protein (Protein Mixture) | Arm 13: ReVacc Subcohort 1C: Ad26.RSV.preF/RSV preF Protein (Protein Mixture) | Arm 14: ReVacc Subcohort 2C: Placebo to Ad26.RSV.preF/RSV preF Protein (Protein Mixture)
Started | 0 | 0 | 120 | 126 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 94 | 102 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 26 | 24 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Site terminated by Sponsor | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 21 | 18 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Revacc Subcohorts (From Day 730 to 1095)
Arm/Group | Arm 1: Main Cohort: Group 1: Ad26.RSV.preF and RSV preF Protein (Protein Mixture) | Arm 2: Main Cohort: Group 2: Placebo | Arm 3: Revaccination (ReVacc) Subcohort 1A: Ad26.RSV.preF/RSV preF Protein (Protein Mixture) | Arm 4: ReVacc Subcohort 2A: Placebo to Ad26.RSV.preF/RSV preF Protein Mixture | Arm 5: ReVacc Subcohort 2A: Placebo to Ad26.RSV.preF/RSV preF Protein + Ad26.RSV.PreF Alone | Arm 6: ReVacc Subcohort 2A: Placebo to Ad26.RSV.preF/RSV preF Protein + RSV preF Protein Alone | Arm 7: ReVacc Subcohort 2A: Placebo to Ad26.RSV.preF/RSV preF Protein (Protein Mixture) | Arm 8: ReVacc Subcohort 1B: Ad26.RSV.preF/RSV preF Protein (Protein Mixture) | Arm 9: ReVacc Subcohort 2B:Placebo to Ad26.RSV.preF/RSV preF Protein (Protein Mixture) | Arm 10: ReVacc Subcohort 2B: Placebo to Ad26.RSV.preF/RSV preF Protein + Ad26.RSV.preF | Arm 11: ReVacc Subcohort 2B: Placebo to Ad26.RSV.preF/RSV preF Protein + RSV preF Protein Alone | Arm 12: ReVacc Subcohort 2B: Placebo to Ad26.RSV.preF/RSV preF Protein (Protein Mixture) | Arm 13: ReVacc Subcohort 1C: Ad26.RSV.preF/RSV preF Protein (Protein Mixture) | Arm 14: ReVacc Subcohort 2C: Placebo to Ad26.RSV.preF/RSV preF Protein (Protein Mixture)
Started | 0 | 0 | 0 | 0 | 28 | 28 | 28 | 137 | 149 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 28 | 24 | 28 | 127 | 3 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 10 | 146 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 0 | 0
Not completed — Study Terminated by Sponsor | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 107 | 0 | 0 | 0 | 0 | 0
Not completed — Site terminated by Sponsor | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 7 | 20 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 4 | 0 | 0 | 0 | 0 | 0
Period: Revacc Subcohort (From Day 1095 to 1460)
Arm/Group | Arm 1: Main Cohort: Group 1: Ad26.RSV.preF and RSV preF Protein (Protein Mixture) | Arm 2: Main Cohort: Group 2: Placebo | Arm 3: Revaccination (ReVacc) Subcohort 1A: Ad26.RSV.preF/RSV preF Protein (Protein Mixture) | Arm 4: ReVacc Subcohort 2A: Placebo to Ad26.RSV.preF/RSV preF Protein Mixture | Arm 5: ReVacc Subcohort 2A: Placebo to Ad26.RSV.preF/RSV preF Protein + Ad26.RSV.PreF Alone | Arm 6: ReVacc Subcohort 2A: Placebo to Ad26.RSV.preF/RSV preF Protein + RSV preF Protein Alone | Arm 7: ReVacc Subcohort 2A: Placebo to Ad26.RSV.preF/RSV preF Protein (Protein Mixture) | Arm 8: ReVacc Subcohort 1B: Ad26.RSV.preF/RSV preF Protein (Protein Mixture) | Arm 9: ReVacc Subcohort 2B:Placebo to Ad26.RSV.preF/RSV preF Protein (Protein Mixture) | Arm 10: ReVacc Subcohort 2B: Placebo to Ad26.RSV.preF/RSV preF Protein + Ad26.RSV.preF | Arm 11: ReVacc Subcohort 2B: Placebo to Ad26.RSV.preF/RSV preF Protein + RSV preF Protein Alone | Arm 12: ReVacc Subcohort 2B: Placebo to Ad26.RSV.preF/RSV preF Protein (Protein Mixture) | Arm 13: ReVacc Subcohort 1C: Ad26.RSV.preF/RSV preF Protein (Protein Mixture) | Arm 14: ReVacc Subcohort 2C: Placebo to Ad26.RSV.preF/RSV preF Protein (Protein Mixture)
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 37 | 37 | 37 | 131 | 119
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 37 | 37 | 37 | 131 | 119
Not completed — Study Terminated by Sponsor | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 36 | 36 | 35 | 125 | 114
Not completed — Site terminated by Sponsor | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 4 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) included all randomized participants with a documented vaccine administration, regardless of the occurrence of protocol deviations.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Main Cohort: Group 1: Ad26.RSV.preF and RSV preF Protein (Protein Mixture) | Arm 2: Main Cohort: Group 2: Placebo | Total
Number analyzed (Participants) | 2891 | 2891 | 5782
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.7 (5.37) | 71.6 (5.38) | 71.7 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1639 | 1694 | 3333
  Male | 1252 | 1197 | 2449
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 85 | 97 | 182
  Not Hispanic or Latino | 2778 | 2773 | 5551
  Unknown or Not Reported | 28 | 21 | 49
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 8 | 9 | 17
  Asian | 15 | 17 | 32
  Native Hawaiian or Other Pacific Islander | 16 | 5 | 21
  Black or African American | 169 | 148 | 317
  White | 2658 | 2690 | 5348
  More than one race | 9 | 14 | 23
  Unknown or Not Reported | 16 | 8 | 24
Region of Enrollment [Count of Participants; unit: Participants]
  UNITED STATES | 2891 | 2891 | 5782

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With First Occurrence of Reverse Transcriptase Polymerase Chain Reaction (RT-PCR)-Confirmed Respiratory Syncytial Virus (RSV) Mediated Lower Respiratory Tract Disease (LRTD)
Description: Number of participants with first occurrence of RT-PCR-confirmed RSV mediated LRTD according to case definition-1, 2 and 3 were reported. Case definition 1 was defined as having a new onset or worsening in 3 or more symptoms of lower respiratory tract infection (LRTI) ; Case definition 2 was defined as having a new onset or worsening in greater than or equal to (>=) 2 symptoms of LRTI; and Case definition 3 was defined as having a new onset or worsening in >=2 OR >=1 symptoms of LRTI with >=1 systemic symptoms. Systemic symptoms (fatigue/malaise and fever/feverishness) and symptoms of LRTI (cough, shortness of breath, sputum production, wheezing and tachypnea) were collected via the RiiQ. RiiQ symptom scale was a 13-items questionnaire rated on a 4-point scale. Each symptom was rated on a scale of 0 to 3 where 0=None, 1=Mild, 2=Moderate, and 3=Severe. Higher scores indicated greater severity. The total LRTD symptom score was calculated as the mean of the LRTD symptom scores.
Time Frame: From screening (Day 1) up to 9 months
Population: The Per-protocol Efficacy (PPE) population included all randomized and vaccinated participants excluding participants with major protocol deviations expecting to impact the efficacy outcomes. Any participant with an RT-PCR-confirmed RSV-mediated acute respiratory infection (ARI) with onset within 14 days after vaccination and participants who discontinued within 14 days after vaccination were excluded from the PPE population.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Main Cohort: Group 1: Ad26.RSV.preF and RSV preF Protein (Protein Mixture) | Arm 2: Main Cohort: Group 2: Placebo
Number analyzed (Participants) | 2791 | 2801
Participants
  Case Definition-1 | 6 | 30
  Case Definition-2 | 10 | 40
  Case Definition-3 | 13 | 43
Statistical Analysis 1: Comparison: Arm 1: Main Cohort: Group 1: Ad26.RSV.preF and RSV preF Protein (Protein Mixture) vs Arm 2: Main Cohort: Group 2: Placebo; Case Definition 1; Test type: Superiority; p = 0.00004, Poisson regression; Event Rate = 80.0, 94.211% CI 2-sided [52.2 to 92.9]
Statistical Analysis 2: Comparison: Arm 1: Main Cohort: Group 1: Ad26.RSV.preF and RSV preF Protein (Protein Mixture) vs Arm 2: Main Cohort: Group 2: Placebo; Case Definition 2; Test type: Superiority; p = 0.00001, Poisson regression; Event Rate = 75.0, 94.211% CI 2-sided [50.1 to 88.5]
Statistical Analysis 3: Comparison: Arm 1: Main Cohort: Group 1: Ad26.RSV.preF and RSV preF Protein (Protein Mixture) vs Arm 2: Main Cohort: Group 2: Placebo; Case Definition 3; Test type: Superiority; p = 0.00004, Poisson regression; Event Rate = 69.8, 94.211% CI 2-sided [43.7 to 84.7]

2. Secondary Outcome: Main Cohorts: Number of Participants With Any RT-PCR-confirmed RSV Disease
Description: Number of participants with any RT-PCR-confirmed RSV disease were reported. The analysis was based on poisson regression model.
Time Frame: From screening (Day 1) up to 9 months
Population: The PPE population included all randomized and vaccinated participants excluding participants with major protocol deviations expecting to impact the efficacy outcomes. Any participant with an RT-PCR-confirmed RSV-mediated ARI with onset within 14 days after vaccination and participants who discontinued within 14 days after vaccination were excluded from the PPE population.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Main Cohort: Group 1: Ad26.RSV.preF and RSV preF Protein (Protein Mixture) | Arm 2: Main Cohort: Group 2: Placebo
Number analyzed (Participants) | 2791 | 2801
Participants | 13 | 43

3. Secondary Outcome: Main Cohorts: Respiratory Syncytial Virus (RSV) A2 Strain Neutralization Antibody Titers
Description: RSV A2 strain neutralizing antibody titers of the vaccine-induced immune response was assessed through virus neutralization assay.
Time Frame: Days 15, 85, 169, 365
Population: Per-protocol Immunogenicity (PPI) population included all randomized and vaccinated participants who were part of the immunogenicity subset and for whom immunogenicity data were available. Here, 'N' (number of participants analyzed) signifies participants who were evaluable for this outcome measure and 'n' (participants analyzed) signifies the participants evaluable at specified timepoints.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Arm 1: Main Cohort: Group 1: Ad26.RSV.preF and RSV preF Protein (Protein Mixture) | Arm 2: Main Cohort: Group 2: Placebo
Number analyzed (Participants) | 95 | 96
Titers
  Day 15: number analyzed (Participants) | 95 | 91
  Day 15 | 6761 [5478 to 8346] | 516 [443 to 602]
  Day 85: number analyzed (Participants) | 94 | 96
  Day 85 | 4963 [4053 to 6077] | 602 [528 to 687]
  Day 169: number analyzed (Participants) | 94 | 93
  Day 169 | 3057 [2523 to 3703] | 552 [489 to 623]
  Day 365: number analyzed (Participants) | 81 | 72
  Day 365 | 1546 [1235 to 1936] | 341 [284 to 409]

4. Secondary Outcome: Revaccination Subcohorts: Respiratory Syncytial Virus (RSV) A2 Strain Neutralization Antibody Titers
Description: as for outcome 3
Time Frame: Days 15, 365, 379, 393, 449, 730, 737, 744, 758
Population: PPI set: all randomized and vaccinated participants who were part of immunogenicity subset and for whom immunogenicity data were available. 'N' (number of participants analyzed): participants evaluable for this outcome measure, 'n' (participants analyzed): participants evaluable at specified timepoints and 'n (number analyzed)=0' signifies that none of participants were available for the assessment at specified timepoints. This outcome measure was planned to be analyzed for specified arms only.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Arm 3: Revaccination (ReVacc) Subcohort 1A: Ad26.RSV.preF/RSV preF Protein (Protein Mixture) | Arm 4: ReVacc Subcohort 2A: Placebo to Ad26.RSV.preF/RSV preF Protein Mixture | Arm 5: ReVacc Subcohort 2A: Placebo to Ad26.RSV.preF/RSV preF Protein + Ad26.RSV.PreF Alone | Arm 6: ReVacc Subcohort 2A: Placebo to Ad26.RSV.preF/RSV preF Protein + RSV preF Protein Alone | Arm 7: ReVacc Subcohort 2A: Placebo to Ad26.RSV.preF/RSV preF Protein (Protein Mixture)
Number analyzed (Participants) | 117 | 120 | 26 | 28 | 27
Titers
  Day 15: number analyzed (Participants) | 111 | 116 | 26 | 24 | 27
  Day 15 | 5508 [4695 to 6460] | 421 [374 to 475] | 357 [281 to 454] | 361 [291 to 448] | 487 [383 to 620]
  Day 365: number analyzed (Participants) | 117 | 120 | 25 | 28 | 27
  Day 365 | 1451 [1275 to 1651] | 402 [354 to 456] | 308 [241 to 392] | 342 [264 to 444] | 435 [348 to 544]
  Day 379: number analyzed (Participants) | 90 | 100 | 23 | 24 | 20
  Day 379 | 2075 [1779 to 2420] | 5416 [4462 to 6573] | 4289 [2739 to 6717] | 6117 [4194 to 8922] | 5114 [3161 to 8275]
  Day 393: number analyzed (Participants) | 97 | 99 | 22 | 20 | 24
  Day 393 | 2098 [1760 to 2501] | 4821 [3982 to 5836] | 4487 [3200 to 6291] | 5008 [3272 to 7664] | 4078 [2524 to 6589]
  Day 449: number analyzed (Participants) | 109 | 105 | 22 | 24 | 26
  Day 449 | 2491 [2183 to 2841] | 4136 [3483 to 4912] | 3186 [2290 to 4433] | 4194 [3108 to 5659] | 3553 [2557 to 4935]
  Day 730: number analyzed (Participants) | 0 | 76 | 24 | 25 | 25
  Day 730 |  | 2260 [1914 to 2669] | 1795 [1319 to 2443] | 2486 [1827 to 3382] | 2491 [1859 to 3338]
  Day 737: number analyzed (Participants) | 0 | 0 | 21 | 23 | 22
  Day 737 |  |  | 2073 [1415 to 3036] | 2677 [2125 to 3373] | 3116 [2303 to 4215]
  Day 744: number analyzed (Participants) | 0 | 0 | 19 | 19 | 21
  Day 744 |  |  | 2542 [1721 to 3753] | 3115 [2453 to 3954] | 3812 [2772 to 5242]
  Day 758: number analyzed (Participants) | 0 | 0 | 15 | 16 | 21
  Day 758 |  |  | 2263 [1423 to 3598] | 3631 [2601 to 5067] | 3668 [2714 to 4958]

5. Secondary Outcome: Revaccination Subcohorts: Geometric Mean Titers (GMTs) of Prefusion F-protein (Pre-F) A Antibodies as Assessed by Enzyme-linked Immunosorbent Assay (ELISA)
Description: GMTs of preF-A antibodies after the administration of Ad26.RSV.preF-based vaccine as assessed by ELISA were reported.
Time Frame: Day 15: Arms 3 to 7,13 and 14; Days 365, 379, 393, 449, 533: Arms 3 to 7; Day 730: Arms 4 to 7; Days 737, 744, 758: Arms 5 to 7; Day 1095, 1109: Arms 13 and 14
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Arm 3: Revaccination (ReVacc) Subcohort 1A: Ad26.RSV.preF/RSV preF Protein (Protein Mixture) | Arm 4: ReVacc Subcohort 2A: Placebo to Ad26.RSV.preF/RSV preF Protein Mixture | Arm 5: ReVacc Subcohort 2A: Placebo to Ad26.RSV.preF/RSV preF Protein + Ad26.RSV.PreF Alone | Arm 6: ReVacc Subcohort 2A: Placebo to Ad26.RSV.preF/RSV preF Protein + RSV preF Protein Alone | Arm 7: ReVacc Subcohort 2A: Placebo to Ad26.RSV.preF/RSV preF Protein (Protein Mixture) | Arm 13: ReVacc Subcohort 1C: Ad26.RSV.preF/RSV preF Protein (Protein Mixture) | Arm 14: ReVacc Subcohort 2C: Placebo to Ad26.RSV.preF/RSV preF Protein (Protein Mixture)
Number analyzed (Participants) | 117 | 120 | 26 | 28 | 27 | 127 | 114
Titers
  Day 15: number analyzed (Participants) | 111 | 116 | 26 | 24 | 27 | 125 | 112
  Day 15 | 4091 [3540 to 4728] | 301 [269 to 336] | 258 [203 to 328] | 282 [228 to 349] | 391 [307 to 497] | 4195 [3685 to 4776] | 279 [238 to 326]
  Day 365: number analyzed (Participants) | 117 | 120 | 25 | 28 | 27 | 0 | 0
  Day 365 | 1003 [901 to 1117] | 325 [293 to 361] | 259 [200 to 335] | 317 [259 to 388] | 358 [291 to 440] |  |
  Day 379: number analyzed (Participants) | 90 | 100 | 23 | 24 | 20 | 0 | 0
  Day 379 | 1688 [1487 to 1917] | 4402 [3807 to 5089] | 3642 [2582 to 5136] | 4827 [3545 to 6572] | 4290 [3069 to 5996] |  |
  Day 393: number analyzed (Participants) | 97 | 99 | 22 | 20 | 24 | 0 | 0
  Day 393 | 1757 [1549 to 1994] | 3793 [3265 to 4405] | 3408 [2578 to 4505] | 4341 [3072 to 6134] | 3541 [2473 to 5070] |  |
  Day 449: number analyzed (Participants) | 109 | 105 | 22 | 24 | 26 | 0 | 0
  Day 449 | 1534 [1376 to 1710] | 2513 [2172 to 2908] | 2227 [1671 to 2968] | 2999 [2254 to 3991] | 2129 [1509 to 3002] |  |
  Day 533: number analyzed (Participants) | 95 | 99 | 20 | 24 | 25 | 0 | 0
  Day 533 | 1430 [1287 to 1590] | 1818 [1585 to 2086] | 1605 [1132 to 2275] | 1835 [1429 to 2358] | 1783 [1350 to 2355] |  |
  Day 730: number analyzed (Participants) | 0 | 75 | 24 | 25 | 25 | 0 | 0
  Day 730 |  | 1270 [1112 to 1451] | 992 [767 to 1283] | 1467 [1182 to 1822] | 1379 [1099 to 1732] |  |
  Day 737: number analyzed (Participants) | 0 | 0 | 21 | 23 | 22 | 0 | 0
  Day 737 |  |  | 1138 [850 to 1524] | 1779 [1510 to 2096] | 1674 [1348 to 2077] |  |
  Day 744: number analyzed (Participants) | 0 | 0 | 19 | 19 | 21 | 0 | 0
  Day 744 |  |  | 1352 [1111 to 1644] | 2001 [1619 to 2473] | 2181 [1714 to 2774] |  |
  Day 758: number analyzed (Participants) | 0 | 0 | 15 | 16 | 21 | 0 | 0
  Day 758 |  |  | 1436 [1049 to 1964] | 2331 [1786 to 3043] | 2131 [1666 to 2726] |  |
  Day 1095: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 127 | 114
  Day 1095 |  |  |  |  |  | 825 [743 to 917] | 317 [276 to 363]
  Day 1109: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 108 | 96
  Day 1109 |  |  |  |  |  | 2152 [1923 to 2407] | 3736 [3196 to 4367]

6. Secondary Outcome: Revaccination Subcohort 2A: T-cell Interferon (IFN) Gamma Responses to RSV F Protein Peptides Analyzed by Enzyme-linked Immunospot Assay (ELISpot)
Description: T-cell IFN gamma responses to RSV F protein specific peptides as measured by ELISpot assay were reported. RSV F protein specific T-cell IFN gamma ELISpot responses were measured as counts of spot forming cells per million peripheral blood mononuclear cells (SFC/10^6 PBMCs).
Time Frame: Days 730, 744, 758
Population: PPI population included all randomized and vaccinated participants who were part of the immuno subset and for whom immunogenicity data were available. Here, 'N' (Overall number of participants analyzed) signifies participants who were evaluable for this outcome measure. Here, 'n' signifies participants evaluable for specified timepoints. This outcome measure was planned to be analyzed for specified arms only.
Measure: Median (Full Range); unit: SFC/10^6 PBMCs
Arm/Group | Arm 5: ReVacc Subcohort 2A: Placebo to Ad26.RSV.preF/RSV preF Protein + Ad26.RSV.PreF Alone | Arm 6: ReVacc Subcohort 2A: Placebo to Ad26.RSV.preF/RSV preF Protein + RSV preF Protein Alone | Arm 7: ReVacc Subcohort 2A: Placebo to Ad26.RSV.preF/RSV preF Protein (Protein Mixture)
Number analyzed (Participants) | 12 | 24 | 16
SFC/10^6 PBMCs
  Day 730 | 129 [34 to 320] | 198 [34 to 1035] | 168 [34 to 795]
  Day 744: number analyzed (Participants) | 11 | 18 | 15
  Day 744 | 402 [105 to 1420] | 498 [130 to 2269] | 405 [34 to 3104]
  Day 758: number analyzed (Participants) | 8 | 12 | 12
  Day 758 | 278 [84 to 443] | 484 [196 to 1375] | 277 [34 to 1253]

7. Secondary Outcome: Main Cohorts: T-cell Interferon (IFN) Gamma Responses to RSV F Protein Peptides Analyzed by Enzyme-linked Immunospot Assay (ELISpot)
Description: as for outcome 6
Time Frame: Days 15, 85, 169, 365, 533
Population: PPI population included all randomized and vaccinated participants who were part of the immuno subset and for whom immunogenicity data were available. Here, 'N' (number of participants analyzed) signifies participants who were evaluable for this outcome measure. Here, 'n' signifies participants evaluable for specified timepoints.
Measure: Median (Full Range); unit: SFC/10^6 PBMCs
Arm/Group | Arm 1: Main Cohort: Group 1: Ad26.RSV.preF and RSV preF Protein (Protein Mixture) | Arm 2: Main Cohort: Group 2: Placebo
Number analyzed (Participants) | 91 | 87
SFC/10^6 PBMCs
  Day 15: number analyzed (Participants) | 76 | 76
  Day 15 | 444 [279 to 641] | 34 [34 to 34]
  Day 85: number analyzed (Participants) | 90 | 87
  Day 85 | 274 [173 to 471] | 34 [34 to 34]
  Day 169 | 201 [123 to 324] | 34 [34 to 34]
  Day 365: number analyzed (Participants) | 75 | 66
  Day 365 | 182 [110 to 297] | 34 [34 to 34]
  Day 533: number analyzed (Participants) | 59 | 56
  Day 533 | 143 [96 to 238] | 34 [34 to 74]

8. Secondary Outcome: Main Cohorts: Number of Participants With Solicited Local Adverse Events (AEs) up to 7 Days After First Vaccination
Description: An AE was any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the intervention. Solicited local AEs were precisely defined events that participants were specifically asked about and which were noted by participants in the diary. Solicited local AEs included erythema, swelling/induration, and pain/tenderness. Per protocol, all solicited local AEs were considered as related to intervention.
Time Frame: Up to Day 8 (7 days after first vaccination on Day 1)
Population: The safety subset included all participants that consented to the collection of AEs (solicited AEs for up to 7 days after vaccination and unsolicited AEs for 28 days after vaccination). Here, 'N' (number of participants analyzed) signifies participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Main Cohort: Group 1: Ad26.RSV.preF and RSV preF Protein (Protein Mixture) | Arm 2: Main Cohort: Group 2: Placebo
Number analyzed (Participants) | 341 | 334
Participants | 132 | 29

9. Secondary Outcome: Main Cohorts: Number of Participants With Solicited Systemic AEs up to 7 Days After First Vaccination
Description: An AE was any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the intervention. Solicited systemic AEs included fatigue, headache, myalgia, arthralgia, and fever (defined as an endogenous elevation of body temperature >=38.0°C, as recorded in at least one measurement).
Time Frame: Up to Day 8 (7 days after first vaccination on Day 1)
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Main Cohort: Group 1: Ad26.RSV.preF and RSV preF Protein (Protein Mixture) | Arm 2: Main Cohort: Group 2: Placebo
Number analyzed (Participants) | 341 | 334
Participants | 143 | 58

10. Secondary Outcome: Main Cohorts: Number of Participants With Unsolicited AEs up to 28 Days After First Vaccination
Description: An AE was any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the intervention. Unsolicited adverse events included all adverse events for which the participant is not specifically questioned in the participant diary.
Time Frame: Up to Day 29 (28 days after first vaccination on Day 1)
Population: The safety subset included all participants that consented to the collection of AEs (solicited AEs for up to 7 days after vaccination and unsolicited AEs for 28 days after vaccination).
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Main Cohort: Group 1: Ad26.RSV.preF and RSV preF Protein (Protein Mixture) | Arm 2: Main Cohort: Group 2: Placebo
Number analyzed (Participants) | 348 | 347
Participants | 58 | 50

11. Secondary Outcome: Revaccination Subcohorts: Number of Participants With Solicited Local AEs 7 Days After Re-vaccination up to 1, 2 and 3 Years
Description: Number of participants with solicited local AEs 7 days after re-vaccination at 1, 2 and 3 years were reported. An AE was any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the intervention. Solicited local AEs were precisely defined events that participants were specifically asked about and which were noted by participants in the diary. Solicited local AEs included erythema, swelling/induration, and pain/tenderness. Per protocol, all solicited local AEs were considered as related to intervention.
Time Frame: Arms 3,4: 7 days after revacc at 1 year (up to Day 372); Arm 5,6,7,8,9: 7 days after revacc at 2 years (up to Day 737); Arms 10,11,12,13,14: 7 days after revacc at 3 year (up to Day 1102)
Population: The Full Analysis Set (FAS) included all randomized participants with a documented vaccine administration, regardless of the occurrence of protocol deviations. Here, 'N' (number of participants analyzed) signifies participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 3: Revaccination (ReVacc) Subcohort 1A: Ad26.RSV.preF/RSV preF Protein (Protein Mixture) | Arm 4: ReVacc Subcohort 2A: Placebo to Ad26.RSV.preF/RSV preF Protein Mixture | Arm 5: ReVacc Subcohort 2A: Placebo to Ad26.RSV.preF/RSV preF Protein + Ad26.RSV.PreF Alone | Arm 6: ReVacc Subcohort 2A: Placebo to Ad26.RSV.preF/RSV preF Protein + RSV preF Protein Alone | Arm 7: ReVacc Subcohort 2A: Placebo to Ad26.RSV.preF/RSV preF Protein (Protein Mixture) | Arm 8: ReVacc Subcohort 1B: Ad26.RSV.preF/RSV preF Protein (Protein Mixture) | Arm 9: ReVacc Subcohort 2B:Placebo to Ad26.RSV.preF/RSV preF Protein (Protein Mixture) | Arm 10: ReVacc Subcohort 2B: Placebo to Ad26.RSV.preF/RSV preF Protein + Ad26.RSV.preF | Arm 11: ReVacc Subcohort 2B: Placebo to Ad26.RSV.preF/RSV preF Protein + RSV preF Protein Alone | Arm 12: ReVacc Subcohort 2B: Placebo to Ad26.RSV.preF/RSV preF Protein (Protein Mixture) | Arm 13: ReVacc Subcohort 1C: Ad26.RSV.preF/RSV preF Protein (Protein Mixture) | Arm 14: ReVacc Subcohort 2C: Placebo to Ad26.RSV.preF/RSV preF Protein (Protein Mixture)
Number analyzed (Participants) | 119 | 126 | 28 | 27 | 28 | 137 | 149 | 37 | 36 | 37 | 131 | 118
Participants | 37 | 31 | 9 | 18 | 12 | 97 | 81 | 26 | 17 | 29 | 93 | 64

12. Secondary Outcome: Revaccination Subcohorts: Number of Participants With Solicited Systemic AEs 7 Days After Re-vaccination up to 1, 2 and 3 Years
Description: Number of participants with solicited systemic AEs 7 days after re-vaccination up to 1, 2 and 3 years were reported. An AE was any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the intervention. Solicited systemic AEs included fatigue, headache, myalgia, arthralgia, and fever (defined as an endogenous elevation of body temperature >=38.0°C, as recorded in at least one measurement).
Time Frame: as for outcome 11
Population: The FAS included all randomized participants with a documented vaccine administration, regardless of the occurrence of protocol deviations. Here, 'N' (number of participants analyzed) signifies participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 3: Revaccination (ReVacc) Subcohort 1A: Ad26.RSV.preF/RSV preF Protein (Protein Mixture) | Arm 4: ReVacc Subcohort 2A: Placebo to Ad26.RSV.preF/RSV preF Protein Mixture | Arm 5: ReVacc Subcohort 2A: Placebo to Ad26.RSV.preF/RSV preF Protein + Ad26.RSV.PreF Alone | Arm 6: ReVacc Subcohort 2A: Placebo to Ad26.RSV.preF/RSV preF Protein + RSV preF Protein Alone | Arm 7: ReVacc Subcohort 2A: Placebo to Ad26.RSV.preF/RSV preF Protein (Protein Mixture) | Arm 8: ReVacc Subcohort 1B: Ad26.RSV.preF/RSV preF Protein (Protein Mixture) | Arm 9: ReVacc Subcohort 2B:Placebo to Ad26.RSV.preF/RSV preF Protein (Protein Mixture) | Arm 10: ReVacc Subcohort 2B: Placebo to Ad26.RSV.preF/RSV preF Protein + Ad26.RSV.preF | Arm 11: ReVacc Subcohort 2B: Placebo to Ad26.RSV.preF/RSV preF Protein + RSV preF Protein Alone | Arm 12: ReVacc Subcohort 2B: Placebo to Ad26.RSV.preF/RSV preF Protein (Protein Mixture) | Arm 13: ReVacc Subcohort 1C: Ad26.RSV.preF/RSV preF Protein (Protein Mixture) | Arm 14: ReVacc Subcohort 2C: Placebo to Ad26.RSV.preF/RSV preF Protein (Protein Mixture)
Number analyzed (Participants) | 119 | 126 | 28 | 27 | 28 | 137 | 149 | 37 | 36 | 37 | 131 | 118
Participants | 35 | 36 | 7 | 15 | 10 | 79 | 85 | 16 | 12 | 25 | 80 | 70

13. Secondary Outcome: Revaccination Subcohorts: Number of Participants With Unsolicited AEs 28 Days After Re-vaccination up to 1, 2 and 3 Years
Description: as for outcome 10
Time Frame: Arms 3,4: 28 days after revacc at 1 year (up to Day 393); Arms 5,6,7,8,9: 28 days after revacc at 2 years (up to Day 758); Arms 10,11,12,13,14: 28 days after revaccination at 3 year (up to Day 1123)
Population: The FAS included all randomized participants with a documented vaccine administration, regardless of the occurrence of protocol deviations.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 3: Revaccination (ReVacc) Subcohort 1A: Ad26.RSV.preF/RSV preF Protein (Protein Mixture) | Arm 4: ReVacc Subcohort 2A: Placebo to Ad26.RSV.preF/RSV preF Protein Mixture | Arm 5: ReVacc Subcohort 2A: Placebo to Ad26.RSV.preF/RSV preF Protein + Ad26.RSV.PreF Alone | Arm 6: ReVacc Subcohort 2A: Placebo to Ad26.RSV.preF/RSV preF Protein + RSV preF Protein Alone | Arm 7: ReVacc Subcohort 2A: Placebo to Ad26.RSV.preF/RSV preF Protein (Protein Mixture) | Arm 8: ReVacc Subcohort 1B: Ad26.RSV.preF/RSV preF Protein (Protein Mixture) | Arm 9: ReVacc Subcohort 2B:Placebo to Ad26.RSV.preF/RSV preF Protein (Protein Mixture) | Arm 10: ReVacc Subcohort 2B: Placebo to Ad26.RSV.preF/RSV preF Protein + Ad26.RSV.preF | Arm 11: ReVacc Subcohort 2B: Placebo to Ad26.RSV.preF/RSV preF Protein + RSV preF Protein Alone | Arm 12: ReVacc Subcohort 2B: Placebo to Ad26.RSV.preF/RSV preF Protein (Protein Mixture) | Arm 13: ReVacc Subcohort 1C: Ad26.RSV.preF/RSV preF Protein (Protein Mixture) | Arm 14: ReVacc Subcohort 2C: Placebo to Ad26.RSV.preF/RSV preF Protein (Protein Mixture)
Number analyzed (Participants) | 120 | 126 | 28 | 28 | 28 | 137 | 149 | 37 | 37 | 37 | 131 | 119
Participants | 6 | 10 | 4 | 5 | 8 | 12 | 16 | 4 | 3 | 4 | 11 | 10

14. Secondary Outcome: Revaccination Subcohorts: Number of Participants With Adverse Events of Special Interests (AESI)
Description: Number of participants with AESIs were reported. An AE was any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Thrombosis with thrombocytopenia syndrome (TTS) was considered as an AESI.
Time Frame: Arms 3,4: 6 months after revacc at 1 year (up to Day 547); Arm 5,6,7,8,9: 6 months after revacc at 2 years (up to Day 912); Arms 10,11,12,13,14: 6 months after revacc at 3 year (up to Day 1277)
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 3: Revaccination (ReVacc) Subcohort 1A: Ad26.RSV.preF/RSV preF Protein (Protein Mixture) | Arm 4: ReVacc Subcohort 2A: Placebo to Ad26.RSV.preF/RSV preF Protein Mixture | Arm 5: ReVacc Subcohort 2A: Placebo to Ad26.RSV.preF/RSV preF Protein + Ad26.RSV.PreF Alone | Arm 6: ReVacc Subcohort 2A: Placebo to Ad26.RSV.preF/RSV preF Protein + RSV preF Protein Alone | Arm 7: ReVacc Subcohort 2A: Placebo to Ad26.RSV.preF/RSV preF Protein (Protein Mixture) | Arm 8: ReVacc Subcohort 1B: Ad26.RSV.preF/RSV preF Protein (Protein Mixture) | Arm 9: ReVacc Subcohort 2B:Placebo to Ad26.RSV.preF/RSV preF Protein (Protein Mixture) | Arm 10: ReVacc Subcohort 2B: Placebo to Ad26.RSV.preF/RSV preF Protein + Ad26.RSV.preF | Arm 11: ReVacc Subcohort 2B: Placebo to Ad26.RSV.preF/RSV preF Protein + RSV preF Protein Alone | Arm 12: ReVacc Subcohort 2B: Placebo to Ad26.RSV.preF/RSV preF Protein (Protein Mixture) | Arm 13: ReVacc Subcohort 1C: Ad26.RSV.preF/RSV preF Protein (Protein Mixture) | Arm 14: ReVacc Subcohort 2C: Placebo to Ad26.RSV.preF/RSV preF Protein (Protein Mixture)
Number analyzed (Participants) | 120 | 126 | 28 | 28 | 28 | 137 | 149 | 37 | 37 | 37 | 131 | 119
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

15. Secondary Outcome: Main Cohorts:Number of Participants With Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. An SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly/birth defect; suspected transmission of any infectious agent via a medicinal product or medically important. For participants who were not revaccinated only SAEs associated with ARIs and complications related to ARIs that classify as SAEs, SAEs classified as related, SAEs resulting in death, and (S)AEs resulting in study discontinuation or from procedures and non-investigational (concomitant) Janssen products were collected.
Time Frame: From Day 1 up to Day 1095
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Main Cohort: Group 1: Ad26.RSV.preF and RSV preF Protein (Protein Mixture) | Arm 2: Main Cohort: Group 2: Placebo
Number analyzed (Participants) | 2891 | 2891
Participants | 203 | 196

16. Secondary Outcome: Revaccination Subcohorts: Number of Participants With Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. An SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly/birth defect; suspected transmission of any infectious agent via a medicinal product or medically important.
Time Frame: as for outcome 14
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 3: Revaccination (ReVacc) Subcohort 1A: Ad26.RSV.preF/RSV preF Protein (Protein Mixture) | Arm 4: ReVacc Subcohort 2A: Placebo to Ad26.RSV.preF/RSV preF Protein Mixture | Arm 5: ReVacc Subcohort 2A: Placebo to Ad26.RSV.preF/RSV preF Protein + Ad26.RSV.PreF Alone | Arm 6: ReVacc Subcohort 2A: Placebo to Ad26.RSV.preF/RSV preF Protein + RSV preF Protein Alone | Arm 7: ReVacc Subcohort 2A: Placebo to Ad26.RSV.preF/RSV preF Protein (Protein Mixture) | Arm 8: ReVacc Subcohort 1B: Ad26.RSV.preF/RSV preF Protein (Protein Mixture) | Arm 9: ReVacc Subcohort 2B:Placebo to Ad26.RSV.preF/RSV preF Protein (Protein Mixture) | Arm 10: ReVacc Subcohort 2B: Placebo to Ad26.RSV.preF/RSV preF Protein + Ad26.RSV.preF | Arm 11: ReVacc Subcohort 2B: Placebo to Ad26.RSV.preF/RSV preF Protein + RSV preF Protein Alone | Arm 12: ReVacc Subcohort 2B: Placebo to Ad26.RSV.preF/RSV preF Protein (Protein Mixture) | Arm 13: ReVacc Subcohort 1C: Ad26.RSV.preF/RSV preF Protein (Protein Mixture) | Arm 14: ReVacc Subcohort 2C: Placebo to Ad26.RSV.preF/RSV preF Protein (Protein Mixture)
Number analyzed (Participants) | 120 | 126 | 28 | 28 | 28 | 137 | 149 | 37 | 37 | 37 | 131 | 119
Participants | 2 | 6 | 0 | 3 | 1 | 4 | 6 | 2 | 0 | 0 | 2 | 2

17. Secondary Outcome: Main Cohorts: Geometric Mean Titers (GMTs) of Prefusion F-protein (Pre-F) A Antibodies as Assessed by Enzyme-linked Immunosorbent Assay (ELISA)
Description: GMTs of preF-A antibodies after the administration of Ad26.RSV.preF-based vaccine as assessed by ELISA were reported.
Time Frame: Days 15, 85, 169, 365, 533
Population: PPI: all randomized and vaccinated participants who were part of immunogenicity subset and for whom immunogenicity data were available. Here, 'N' (Overall number of participants analyzed)=participants who were evaluable for this outcome measure, "n"=participants evaluable for specific timepoints.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Arm 1: Main Cohort: Group 1: Ad26.RSV.preF and RSV preF Protein (Protein Mixture) | Arm 2: Main Cohort: Group 2: Placebo
Number analyzed (Participants) | 95 | 96
Titers
  Day 15: number analyzed (Participants) | 95 | 91
  Day 15 | 4001 [3354 to 4772] | 305 [256 to 364]
  Day 85: number analyzed (Participants) | 94 | 96
  Day 85 | 2475 [2129 to 2876] | 359 [302 to 426]
  Day 169: number analyzed (Participants) | 94 | 93
  Day 169 | 1604 [1381 to 1863] | 335 [293 to 383]
  Day 365: number analyzed (Participants) | 81 | 72
  Day 365 | 1044 [908 to 1201] | 281 [237 to 334]
  Day 533: number analyzed (Participants) | 70 | 63
  Day 533 | 991 [863 to 1137] | 315 [267 to 371]

ADVERSE EVENTS:
Time Frame: All-cause mortality: Day 1 to Day 1095 (Arms 1, 2); Day 365 to Day 730 (Arms 3, 4); Day 730 to Day 1095 (Arms 5 to 9); Day 1095 to Day 1460 (Arms 10 to 14); Serious/other AEs: Day 1 to Day 1095 (Arms 1, 2), 6 months after revacc at Day 365 (Arms 3, 4): up to Day 547, 6 months after revacc at Day 730 (Arms 5 to 9): up to Day 912, 6 months after revacc at Day 1095 (Arms 10 to 14): up to Day 1277
Description: All-cause mortality and SAEs analyzed based on FAS population which included all randomized participants with a documented vaccine administration, regardless of occurrence of protocol deviations. Other (not including serious) AEs as solicited and unsolicited AEs were collected and analyzed in safety subset (subset of FAS) for main cohorts and in FAS for revaccination subcohorts. The safety subset included all participants that consented to the collection of AEs (solicited and unsolicited AEs).
Arm/Group | Arm 1: Main Cohort: Group 1: Ad26.RSV.preF and RSV preF Protein (Protein Mixture) | Arm 2: Main Cohort: Group 2: Placebo | Arm 3: Revaccination (ReVacc) Subcohort 1A: Ad26.RSV.preF/RSV preF Protein (Protein Mixture) | Arm 4: ReVacc Subcohort 2A: Placebo to Ad26.RSV.preF/RSV preF Protein Mixture | Arm 5: ReVacc Subcohort 2A: Placebo to Ad26.RSV.preF/RSV preF Protein + Ad26.RSV.PreF Alone | Arm 6: ReVacc Subcohort 2A: Placebo to Ad26.RSV.preF/RSV preF Protein + RSV preF Protein Alone | Arm 7: ReVacc Subcohort 2A: Placebo to Ad26.RSV.preF/RSV preF Protein (Protein Mixture) | Arm 8: ReVacc Subcohort 1B: Ad26.RSV.preF/RSV preF Protein (Protein Mixture) | Arm 9: ReVacc Subcohort 2B:Placebo to Ad26.RSV.preF/RSV preF Protein (Protein Mixture) | Arm 10: ReVacc Subcohort 2B: Placebo to Ad26.RSV.preF/RSV preF Protein + Ad26.RSV.preF | Arm 11: ReVacc Subcohort 2B: Placebo to Ad26.RSV.preF/RSV preF Protein + RSV preF Protein Alone | Arm 12: ReVacc Subcohort 2B: Placebo to Ad26.RSV.preF/RSV preF Protein (Protein Mixture) | Arm 13: ReVacc Subcohort 1C: Ad26.RSV.preF/RSV preF Protein (Protein Mixture) | Arm 14: ReVacc Subcohort 2C: Placebo to Ad26.RSV.preF/RSV preF Protein (Protein Mixture)
All-Cause Mortality (participants affected / at risk) | 39/2891 | 38/2891 | 1/120 | 0/126 | 0/28 | 0/28 | 0/28 | 0/137 | 2/149 | 0/37 | 0/37 | 0/37 | 0/131 | 1/119
Serious Adverse Events (participants affected / at risk) | 203/2891 | 196/2891 | 2/120 | 6/126 | 0/28 | 3/28 | 1/28 | 4/137 | 6/149 | 2/37 | 0/37 | 0/37 | 2/131 | 2/119
Other Adverse Events (participants affected / at risk) | 186/348 | 90/347 | 47/120 | 47/126 | 15/28 | 21/28 | 21/28 | 110/137 | 111/149 | 30/37 | 22/37 | 34/37 | 107/131 | 84/119
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: Main Cohort: Group 1: Ad26.RSV.preF and RSV preF Protein (Protein Mixture) (N=2891) | Arm 2: Main Cohort: Group 2: Placebo (N=2891) | Arm 3: Revaccination (ReVacc) Subcohort 1A: Ad26.RSV.preF/RSV preF Protein (Protein Mixture) (N=120) | Arm 4: ReVacc Subcohort 2A: Placebo to Ad26.RSV.preF/RSV preF Protein Mixture (N=126) | Arm 5: ReVacc Subcohort 2A: Placebo to Ad26.RSV.preF/RSV preF Protein + Ad26.RSV.PreF Alone (N=28) | Arm 6: ReVacc Subcohort 2A: Placebo to Ad26.RSV.preF/RSV preF Protein + RSV preF Protein Alone (N=28) | Arm 7: ReVacc Subcohort 2A: Placebo to Ad26.RSV.preF/RSV preF Protein (Protein Mixture) (N=28) | Arm 8: ReVacc Subcohort 1B: Ad26.RSV.preF/RSV preF Protein (Protein Mixture) (N=137) | Arm 9: ReVacc Subcohort 2B:Placebo to Ad26.RSV.preF/RSV preF Protein (Protein Mixture) (N=149) | Arm 10: ReVacc Subcohort 2B: Placebo to Ad26.RSV.preF/RSV preF Protein + Ad26.RSV.preF (N=37) | Arm 11: ReVacc Subcohort 2B: Placebo to Ad26.RSV.preF/RSV preF Protein + RSV preF Protein Alone (N=37) | Arm 12: ReVacc Subcohort 2B: Placebo to Ad26.RSV.preF/RSV preF Protein (Protein Mixture) (N=37) | Arm 13: ReVacc Subcohort 1C: Ad26.RSV.preF/RSV preF Protein (Protein Mixture) (N=131) | Arm 14: ReVacc Subcohort 2C: Placebo to Ad26.RSV.preF/RSV preF Protein (Protein Mixture) (N=119)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood Loss Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Splenic Infarction (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute Coronary Syndrome (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute Left Ventricular Failure (Cardiac disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute Myocardial Infarction (Cardiac disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Angina Unstable (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aortic Valve Disease (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aortic Valve Stenosis (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arteriosclerosis Coronary Artery (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial Fibrillation (Cardiac disorders) | 10 | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial Flutter (Cardiac disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac Arrest (Cardiac disorders) | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac Failure (Cardiac disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac Failure Congestive (Cardiac disorders) | 9 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cardiomyopathy (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Coronary Artery Disease (Cardiac disorders) | 2 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ischaemic Cardiomyopathy (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Left Ventricular Failure (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myocardial Infarction (Cardiac disorders) | 8 | 9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myocardial Ischaemia (Cardiac disorders) | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stress Cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ventricular Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Inappropriate Antidiuretic Hormone Secretion (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Duodenal Ulcer Haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Food Poisoning (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastric Perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hiatus Hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Inguinal Hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intestinal Obstruction (Gastrointestinal disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intestinal Perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Large Intestinal Obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Obstructive Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oesophageal Obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oesophageal Perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatic Cyst (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatic Mass (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatitis Acute (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rectal Prolapse (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Adverse Drug Reaction (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest Discomfort (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest Pain (General disorders) | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Death (General disorders) | 7 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Drowning (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Generalised Oedema (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Multiple Organ Dysfunction Syndrome (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Non-Cardiac Chest Pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cirrhosis Alcoholic (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abscess Neck (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alpha Haemolytic Streptococcal Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Clostridium Difficile Colitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Covid-19 (Infections and infestations) | 13 | 13 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Covid-19 Pneumonia (Infections and infestations) | 13 | 16 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Device Related Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diabetic Foot Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gangrene (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Kidney Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Meningitis Aseptic (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Periorbital Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 16 | 10 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia Aspiration (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia Bacterial (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia Chlamydial (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia Mycoplasmal (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia Parainfluenzae Viral (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Septic Shock (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Streptococcal Sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ankle Fracture (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Carbon Monoxide Poisoning (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cervical Vertebral Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Craniocerebral Injury (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Environmental Exposure (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Extradural Haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Facial Bones Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Femur Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fracture Displacement (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Head Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hip Fracture (Injury, poisoning and procedural complications) | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Humerus Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypobarism (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Post Procedural Complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Scapula Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin Abrasion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Subdural Haematoma (Injury, poisoning and procedural complications) | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tibia Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Traumatic Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper Limb Fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wound Dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Wrist Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Adult Failure to Thrive (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cervical Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chondrocalcinosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Kyphoscoliosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 7 | 6 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute Myeloid Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Adenocarcinoma of Colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bladder Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Brain Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cancer Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Endometrial Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatocellular Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Her2 Positive Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intraductal Proliferative Breast Lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Invasive Ductal Breast Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lung Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lung Carcinoma Cell Type Unspecified Stage Iii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lung Carcinoma Cell Type Unspecified Stage Iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Marginal Zone Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Metastases to Liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Metastatic Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Metastatic Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Non-Hodgkin's Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Non-Small Cell Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oesophageal Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ovarian Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ovarian Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatic Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatic Carcinoma Stage Iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Papillary Serous Endometrial Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Prostate Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Small Cell Lung Cancer Extensive Stage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Throat Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Transitional Cell Cancer of the Renal Pelvis and Ureter (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Uterine Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Waldenstrom's Macroglobulinaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Autonomic Neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Carotid Artery Stenosis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebral Haemorrhage (Nervous system disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebral Ischaemia (Nervous system disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebrovascular Accident (Nervous system disorders) | 2 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intracranial Aneurysm (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ischaemic Stroke (Nervous system disorders) | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lacunar Infarction (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lumbar Radiculopathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Metabolic Encephalopathy (Nervous system disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myelopathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peroneal Nerve Palsy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Subarachnoid Haemorrhage (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Toxic Encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Transient Ischaemic Attack (Nervous system disorders) | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Trigeminal Neuralgia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alcoholism (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bipolar Disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depression Suicidal (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Major Depression (Psychiatric disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mental Status Changes (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute Kidney Injury (Renal and urinary disorders) | 2 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chronic Kidney Disease (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neurogenic Bladder (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal Colic (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal Failure (Renal and urinary disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal Injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Postmenopausal Haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 7 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 10 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary Fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rotator Cuff Repair (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aortic Aneurysm (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aortic Stenosis (Vascular disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arteriosclerosis (Vascular disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Endothelial Dysfunction (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertensive Urgency (Vascular disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral Arterial Occlusive Disease (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral Ischaemia (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vascular Compression (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: Main Cohort: Group 1: Ad26.RSV.preF and RSV preF Protein (Protein Mixture) (N=348) | Arm 2: Main Cohort: Group 2: Placebo (N=347) | Arm 3: Revaccination (ReVacc) Subcohort 1A: Ad26.RSV.preF/RSV preF Protein (Protein Mixture) (N=120) | Arm 4: ReVacc Subcohort 2A: Placebo to Ad26.RSV.preF/RSV preF Protein Mixture (N=126) | Arm 5: ReVacc Subcohort 2A: Placebo to Ad26.RSV.preF/RSV preF Protein + Ad26.RSV.PreF Alone (N=28) | Arm 6: ReVacc Subcohort 2A: Placebo to Ad26.RSV.preF/RSV preF Protein + RSV preF Protein Alone (N=28) | Arm 7: ReVacc Subcohort 2A: Placebo to Ad26.RSV.preF/RSV preF Protein (Protein Mixture) (N=28) | Arm 8: ReVacc Subcohort 1B: Ad26.RSV.preF/RSV preF Protein (Protein Mixture) (N=137) | Arm 9: ReVacc Subcohort 2B:Placebo to Ad26.RSV.preF/RSV preF Protein (Protein Mixture) (N=149) | Arm 10: ReVacc Subcohort 2B: Placebo to Ad26.RSV.preF/RSV preF Protein + Ad26.RSV.preF (N=37) | Arm 11: ReVacc Subcohort 2B: Placebo to Ad26.RSV.preF/RSV preF Protein + RSV preF Protein Alone (N=37) | Arm 12: ReVacc Subcohort 2B: Placebo to Ad26.RSV.preF/RSV preF Protein (Protein Mixture) (N=37) | Arm 13: ReVacc Subcohort 1C: Ad26.RSV.preF/RSV preF Protein (Protein Mixture) (N=131) | Arm 14: ReVacc Subcohort 2C: Placebo to Ad26.RSV.preF/RSV preF Protein (Protein Mixture) (N=119)
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Angina Pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Aortic Valve Incompetence (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial Flutter (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mitral Valve Incompetence (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tricuspid Valve Incompetence (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dental Caries (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Solicited) (Gastrointestinal disorders) | 31 | 7 | 4 | 5 | 0 | 3 | 0 | 10 | 22 | 3 | 1 | 4 | 9 | 12
Plicated Tongue (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fatigue (Solicited) (General disorders) | 95 | 42 | 19 | 24 | 4 | 6 | 13 | 66 | 63 | 13 | 8 | 19 | 61 | 57
Oedema Peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (Solicited) (General disorders) | 15 | 0 | 3 | 4 | 0 | 0 | 2 | 5 | 12 | 0 | 0 | 4 | 8 | 7
Vaccination Site Erythema (Solicited) (General disorders) | 22 | 7 | 8 | 4 | 0 | 1 | 4 | 11 | 6 | 1 | 2 | 4 | 18 | 7
Vaccination Site Pain (Solicited) (General disorders) | 120 | 24 | 37 | 29 | 9 | 11 | 18 | 93 | 81 | 26 | 16 | 29 | 91 | 64
Vaccination Site Swelling (Solicited) (General disorders) | 12 | 6 | 8 | 4 | 0 | 1 | 3 | 10 | 8 | 0 | 3 | 4 | 17 | 4
Candida Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Covid-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Oral Candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Respiratory Tract Infection (Infections and infestations) | 13 | 14 | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 8 | 10 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 2 | 4 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Thermal Burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Upper Limb Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Heart Rate Irregular (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 2 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Myalgia (Solicited) (Musculoskeletal and connective tissue disorders) | 95 | 30 | 18 | 24 | 5 | 4 | 9 | 38 | 51 | 10 | 3 | 14 | 40 | 32
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diabetic Neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 5 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Headache (Solicited) (Nervous system disorders) | 83 | 30 | 21 | 19 | 4 | 4 | 10 | 40 | 47 | 10 | 5 | 7 | 42 | 40
Radicular Pain (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Nasal Polyps (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sleep Apnoea Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth Extraction (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will with hold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2023-02-16): https://cdn.clinicaltrials.gov/large-docs/99/NCT03982199/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-11): https://cdn.clinicaltrials.gov/large-docs/99/NCT03982199/SAP_003.pdf